CLINICAL TRIAL: NCT00579774
Title: Effects of Glycoxidative Stress on Human Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 03-0116; 5R37AG023188 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Aging
Keywords: Aging; oxidative stress; glycoxidative stress; glycation; inflammation; nutrition; low AGE intake; dietary AGEs
MeSH Terms: conditions — Inflammation | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Low AGE Diet (Experimental): Low Age Diet
  Interventions: Other: Low AGE Diet
- 2 - Regular Diet (Active Comparator): Regular Diet
  Interventions: Other: Regular Diet

INTERVENTIONS:
Other: Low AGE Diet — Diet
  Arms: 1 - Low AGE Diet
Other: Regular Diet — Diet
  Arms: 2 - Regular Diet

SUMMARY:
Advanced glycation products or AGEs are a heterogeneous group of molecules formed by exposure of tissue constituents to high levels of reducing sugars, e.g. glucose. The interaction of these compounds with extra- and intra-cellular components may account in part for several conditions related to aging. It has recently been recognized that AGEs are also formed during the preparation of food by heating, are absorbed into the circulation and become largely incorporated into tissue components. Accumulation of these exogenous substances over time may, together with those generated endogenously, contribute to the clinical manifestations and complications of aging.

This is an interventional-randomized study in which we are trying to determine whether a diet low in AGE can effectively reduce circulating AGE levels, with or without altering oxidation or inflammatory markers, in a subset of both young and older subjects , over a period of 4 months. If positive results are obtained, longer-term prospective studies will be designed to determine if this intervention can affect disease outcomes in older age subjects.

The study design is very simple and consists initially of obtaining a dietary history, a blood sample, 24-hour urine collection and, subsequently, of determining the effects of a low-AGE diet for 4 months on the plasma levels of these compounds in a group of healthy subjects.

DETAILED DESCRIPTION:
Advancing age is known to be associated with increased oxidant stress (OS), increased prevalence of cardiovascular disease, impaired glucose tolerance, diabetes mellitus, decline of renal function, and accumulation of advanced glycation end products (AGEs). AGEs can lead to activation of transcriptional pathways, excessive proliferative/growth-related phenomena and sustained inflammation and through these different mechanisms may contribute significantly to the clinical complications of aging. Recently, it has become clear that a major source of AGE precursors and OS is the Western diet. The body turnover of AGEs involves specific receptors and is also dependent on renal function.

While experimental work has linked AGE-mediated OS and chronic complications in aging animals, human studies are strikingly lacking. We plan to test the following two hypotheses: 1) older men and women (age > 60 years) who consume standard diets (usually high in AGE content) will have higher serum levels of AGEs in conjunction with higher markers of OS, vascular dysfunction and inflammation when compared with younger subjects (age < 35 but >18 years), and 2) dietary AGE restriction will reduce the serum levels of AGE, markers of OS, vascular dysfunction and inflammation and attenuate the difference between older and younger groups.

Specific aims:

To determine the effect of dietary AGE modification for 4 months on circulating levels of AGEs, markers of oxidative stress, vascular dysfunction, inflammatory mediators and AGE-receptor mechanisms in PBMN in old and young subjects. This will be a randomized study (Study 2).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects of any gender or race between the ages of 18 and 35 or older than 60 years

Exclusion Criteria:

* Diagnosis of diabetes (absence of diabetes will be defined as a negative history of diabetes in combination with a HgbA1c < 6% at the time of recruitment)
* Any major cardiovascular event (myocardial infarction, stroke, PTCA or coronary artery bypass) within the preceding 3 months
* Smokers
* Glucocorticoid, anticoagulant (except for aspirin) or antioxidant therapy
* Serum creatinine greater than 2 mg/dl
* Inability to understand or unwillingness to follow study diets
* Any severe illness with an expected patient survival less than 1 year
* Patients who have initiated therapy with ACE inhibitors, lipid lowering medications or hormone replacement within the previous 3 months. Patients on stable doses of these medications will be included
* Before randomization all subjects will be screened with a 3-day food record to determine their average spontaneous daily intake of AGEs. Only those subjects whose daily intake is on the upper half of normal (greater than 14 AGE Eq/day) will participate in the study. This value of 14 E/day corresponds to the median daily AGE intake estimated in a large number of healthy subjects.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 438 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Levels of AGE | Monthly

SECONDARY OUTCOMES:
Side Effect Measurement | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Helen Vlassara, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Cai W, Uribarri J, Zhu L, Chen X, Swamy S, Zhao Z, Grosjean F, Simonaro C, Kuchel GA, Schnaider-Beeri M, Woodward M, Striker GE, Vlassara H. Oral glycotoxins are a modifiable cause of dementia and the metabolic syndrome in mice and humans. Proc Natl Acad Sci U S A. 2014 Apr 1;111(13):4940-5. doi: 10.1073/pnas.1316013111. Epub 2014 Feb 24. PMID 24567379
- [Result] Uribarri J, Cai W, Pyzik R, Goodman S, Chen X, Zhu L, Ramdas M, Striker GE, Vlassara H. Suppression of native defense mechanisms, SIRT1 and PPARgamma, by dietary glycoxidants precedes disease in adult humans; relevance to lifestyle-engendered chronic diseases. Amino Acids. 2014 Feb;46(2):301-9. doi: 10.1007/s00726-013-1502-4. Epub 2013 May 1. PMID 23636469
- [Result] Uribarri J, Cai W, Ramdas M, Goodman S, Pyzik R, Chen X, Zhu L, Striker GE, Vlassara H. Restriction of advanced glycation end products improves insulin resistance in human type 2 diabetes: potential role of AGER1 and SIRT1. Diabetes Care. 2011 Jul;34(7):1610-6. doi: 10.2337/dc11-0091. PMID 21709297
- [Result] Beeri MS, Moshier E, Schmeidler J, Godbold J, Uribarri J, Reddy S, Sano M, Grossman HT, Cai W, Vlassara H, Silverman JM. Serum concentration of an inflammatory glycotoxin, methylglyoxal, is associated with increased cognitive decline in elderly individuals. Mech Ageing Dev. 2011 Nov-Dec;132(11-12):583-7. doi: 10.1016/j.mad.2011.10.007. Epub 2011 Nov 3. PMID 22079406
- [Result] Vlassara H, Cai W, Goodman S, Pyzik R, Yong A, Chen X, Zhu L, Neade T, Beeri M, Silverman JM, Ferrucci L, Tansman L, Striker GE, Uribarri J. Protection against loss of innate defenses in adulthood by low advanced glycation end products (AGE) intake: role of the antiinflammatory AGE receptor-1. J Clin Endocrinol Metab. 2009 Nov;94(11):4483-91. doi: 10.1210/jc.2009-0089. Epub 2009 Oct 9. PMID 19820033
- [Result] Uribarri J, Woodruff S, Goodman S, Cai W, Chen X, Pyzik R, Yong A, Striker GE, Vlassara H. Advanced glycation end products in foods and a practical guide to their reduction in the diet. J Am Diet Assoc. 2010 Jun;110(6):911-16.e12. doi: 10.1016/j.jada.2010.03.018. PMID 20497781
- [Result] Vlassara H, Uribarri J, Ferrucci L, Cai W, Torreggiani M, Post JB, Zheng F, Striker GE. Identifying advanced glycation end products as a major source of oxidants in aging: implications for the management and/or prevention of reduced renal function in elderly persons. Semin Nephrol. 2009 Nov;29(6):594-603. doi: 10.1016/j.semnephrol.2009.07.013. PMID 20006791